CLINICAL TRIAL: NCT04177641
Title: Investigation of Thiol-disulfide Balance in Cervical Preinvasive Lesions
Brief Title: Evaluation of Thioldisulfide Balance in Cervical Preinvasive Lesions
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: 19/09/2018-15-3
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Oxidative Stress; Low Grade Squamous Intraepithelial Lesion; High-Grade Squamous Intraepithelial Lesions
Keywords: thiol disulfide balance; preinvasive lesion; cervix; oxidative stress
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low grade squamous intraepithelial lesion(LGSIL): low grade squamous intraepithelial lesion(LGSIL) n=100
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L)
- high grade squamous intraepithelial lesion(HGSIL): high grade squamous intraepithelial lesion(HGSIL) n=100
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L)
- Healthy controls: Healthy volunteers n=100
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L)

INTERVENTIONS:
Diagnostic Test: Disulphide(μmol/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with sphectrophotometry
  Other Names: Native thiol (μmol/L); Total thiol (μmol/L); Nativethiol/totalthiol(%); Disulfide/nativethiol(%); Disulfide/totalthiol(%)
Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with sphectrophotometry
  Other Names: Total Antioxidant Capacity(mmolTroloxEquiv/L); Oxidative stress Index (Arbitrary Unite)

SUMMARY:
The purpose of this study is to investigate Thiol-disulfide balance in patients with cervical preinvasive lesions

DETAILED DESCRIPTION:
To date various oxidative stress paramaters were studied in patients with cervical preinvasive lesions, however dynamic thiol disulfide hemostasis has not been previously investigated. The thiol-disulfide balance in the circulation will be measured by the automated system created by Erel & Neselioglu(1).

References 1- Erel O, Neselioglu S. A novel and automated assay for thiol/ disulphide homeostasis. Clin Biochem 2014;47:326-32. doi:10.1016/ j.clinbiochem.2014.09.026.

ELIGIBILITY:
Inclusion Criteria:

• Histopathologically confirmed diagnosis of LGSIL or HGSIL

Exclusion Criteria:

* pulmonary disease
* pulmonary hypertension
* cardiac dysfunction
* renal dysfunction
* liver disease
* chronic ishemia
* systemic inflammation
* other cervical biopy results than LGSIL or HGSIL
* concomitant malignancy
* patients who use vitamin A,C or E (antioxidant vitamins)
* patients who use smoke • patients who use drink alcohol
* patients who use addictive for any drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — histopathologically confirmed LGSIL or HGSIL
Study Population: The diagnosis of preinvasive cervical lesions was made histopathologically by cervical biopsy. An experienced pathologist performed histopathologic examinations
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
serum native thiol level | baseline (preoperative in the morning or preprandial for healthy volunteers)
  serum native thiol level in μmol/L
serum disulphide level | baseline (preoperative in the morning or preprandial for healthy volunteers)
  serum disulphide level in μmol/L
serum total thiol level | baseline (preoperative in the morning or preprandial for healthy volunteers)
  serum total thiol level in μmol/L
the disulphide/native thiol ratio | baseline (preoperative in the morning or preprandial for healthy volunteers)
  the disulphide/native thiol ratio X (100 )
disulphide/total thiol ratio | baseline (preoperative in the morning or preprandial for healthy volunteers)
  disulphide/total thiol ratio X (100 )
native thiol/total thiol ratio | baseline (preoperative in the morning or preprandial for healthy volunteers)
  native thiol/total thiol ratio X (100 )

SECONDARY OUTCOMES:
total antioxidant capacity (TAC) | baseline (preoperative in the morning or preprandial for healthy volunteers)
  TAC in mmol trolox equivalent/L
total oxidant capacity (TOC) | baseline (preoperative in the morning or preprandial for healthy volunteers)
  TOC in mmol H2O2 equivalent/L
Oxidative stress index (OSI) | baseline (preoperative in the morning or preprandial for healthy volunteers)
  OSI in mmol trolox/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)